CLINICAL TRIAL: NCT05380128
Title: Association Study Between Vitamin D Receptor Gene Polymorphisms and Risk and Features of Myasthenia Gravis in Han Chinese Population
Brief Title: Association Study Between VDR Gene Polymorphisms and Risk and Features of MG in Han Chinese Population
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BeijingTH-20220509
Record Dates: First submitted 2022-05-11; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Myasthenia Gravis, Ocular; Gene Polymorphism
MeSH Terms: conditions — Myasthenia Gravis | interventions — Genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MG group: Unrelated patients with MG were included in the study. They were enrolled in the Neurology Department of Beijing Tongren Hospital, Capital Medical University and fulfilled the clinical and electromyography diagnostic criteria for acquired MG. Simply, all MG patients met the following diagnostic criteria: typical symptoms of fluctuating muscle weakness, positive result of neostigmine test, and decremental response to low-frequency repetitive nerve stimulation. Information on age at onset, AChR / MuSK Abs status (partly), thymus status, involved muscles at onset and Osserman type at the maximum worsening during 2 years follow-up were obtained and used as the grouping basis of sub-classifications. They were genotyped for VDR rs1544410, rs2228570, rs731236, and rs7975232 polymorphisms
  Interventions: Genetic: Genotype analysis for VDR rs1544410, rs2228570, rs731236, and rs7975232 polymorphisms
- Healthy control: The geography and ethnically matched control group consisted of 146 unrelated healthy subjects. They were genotyped for VDR rs1544410, rs2228570, rs731236, and rs7975232 polymorphisms.
  Interventions: Genetic: Genotype analysis for VDR rs1544410, rs2228570, rs731236, and rs7975232 polymorphisms

INTERVENTIONS:
Genetic: Genotype analysis for VDR rs1544410, rs2228570, rs731236, and rs7975232 polymorphisms — Genomic DNA was extracted from peripheral blood samples using a Wizard Genomic DNA Purification Kit (Promega, Madison,Wisconsin, USA) as per the product instruction. VDR (rs731236, rs1544410, rs7975232, rs2228570) polymorphisms were genotyped by the improved Multiple Ligase Detection Reaction (iMLDR) developed by Genesky Biotechnologies Inc. (Shanghai, China).

SUMMARY:
The Vitamin D receptor gene (VDR) polymorphisms are the candidate genetic variants for susceptibility to autoimmune diseases. In the present study, the investigators aimed to assess the association between VDR polymorphisms and myasthenia gravis (MG) susceptibility and disease features in Chinese Han population.The patients with MG and healthy controls were genotyped for VDR rs1544410, rs2228570, rs731236, and rs7975232 polymorphisms using the improved multiple ligase detection reaction. Information on age at onset, acetylcholine receptor antibody (AChR-Ab) and muscle-specific kinase antibody (MuSK-Ab) status, thymus status, involved muscles at onset and Osserman type at the maximum worsening during 2 years follow-up were obtained and used as the grouping basis of sub-classifications. Intergroup comparisons of allele and genotype frequencies, haplotype distributions were performed between MG group and the control group, and between each pair of MG subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of myasthenia gravis.
* Han Chinese population.
* Must be able to complete a 2-year follow-up visit.

Exclusion Criteria:

* Clinical data collection can not be completed.
* Poor compliance.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed myasthenia gravis and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Association between VDR gene polymorphism and MG susceptibility | up to 2 years
  Codominant, dominant and recessive genetic models and haplotype analysis were applied to compare the difference between MG and control groups.

SECONDARY OUTCOMES:
Association of VDR gene polymorphism with MG subgroups | up to 2 years
  To study the precise effect of single nucleotide polymorphisms (SNPs) in the different population, the MG patients were divided into subgroups according to essential clinical variables, including onset age (≤50 or >50 years), thymus status (thymoma or non-thymoma, by pathology), AChR / MuSK Abs (positive or negative), onset involvement (ocular or generalized) and Osserman type at the maximum worsening (type I or IIa-IIb or III-V). The investigators analyzed the distribution of genes in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The IPD that support the findings of this study are available from the central contact person upon reasonable request.

REFERENCES:
- [Derived] Dai Y, Wu F, Ni S, Guo S, Lu L, Zhao X. Vitamin D receptor gene polymorphisms are associated with the risk and features of myasthenia gravis in the Han Chinese population. Immunol Res. 2023 Jun;71(3):404-412. doi: 10.1007/s12026-022-09349-x. Epub 2023 Jan 7. PMID 36609978